CLINICAL TRIAL: NCT02915263
Title: A Double-Blind, Randomized, Placebo-Controlled Trial To Evaluate The Efficacy Of Intravenous Immunoglobulin Therapy In Treatment Induced Neuropathy Of Diabetes
Brief Title: The Efficacy Of Intravenous Immunoglobulin Therapy In Treatment Induced Neuropathy Of Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn in the midst of the COVID pandemic
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Christopher Gibbons, MD, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000166
Record Dates: First submitted 2016-08-08; First posted 2016-09-27 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Complications; Diabetes Mellitus; Diabetic Neuropathies
Keywords: Diabetes Complications; Diabetes Mellitus; Diabetic Neuropathies; IGIV-C; Immune Globulin Injection (Human), 10% Caprylate/Chromatography; Gamunex-C
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Diabetic Neuropathies | interventions — Immunoglobulins; Caprylates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.9% Sodium Chloride (Placebo Comparator): The study will include a total 20 individuals. Subjects will be randomized equally to treatment or placebo. The placebo will consist of 0.9% Sodium Chloride per day over 5 days. Participants who are randomized to placebo will receive the same volume as they would if they were randomized to IVIG (i.e.: as if receiving IVIG at 2gm/kg) through a peripheral IV line.
  Interventions: Drug: 0.9% Sodium Chloride
- IGIV-C (Experimental): The study will include a total 20 individuals. Subjects will be randomized equally to treatment or placebo. The treatment will consist of IVIG administered at 2 grams/kg divided over 5 days, with a follow up treatment 3 weeks (+/-3 days) later of IVIG 1gram/kg administered over 2 day (or placebo).
  Interventions: Drug: IGIV-C

INTERVENTIONS:
Drug: IGIV-C — Gamunex-C [immune globulin injection (human) 10% caprylate/chromatography purified] is a sterile solution of human immune globulin protein.
  Other Names: Gamunex-C Liquid; Immune globulin injection (human), 10% caprylate/chromatography purified
  Arms: IGIV-C
Drug: 0.9% Sodium Chloride — Sodium Chloride (also known as saline) is a solution of sodium chloride, or salt, and sterile water.
  Other Names: Saline; 0.9%NaCl
  Arms: 0.9% Sodium Chloride

SUMMARY:
The goal of this pilot study is to obtain preliminary data on the magnitude of the treatment effect of IVIG on the neuropathic pain and neuropathy severity associated with treatment induced neuropathy (TIND).

The investigators hypothesize that immune globulin, administered intravenously (IVIG), will reduce the pain associated with treatment induced neuropathy and reduce the neuropathy severity.

Treatment induced neuropathy in diabetes, is an iatrogenic complications of diabetes. The preliminary data will be used to power a larger treatment trial, and to aid the understanding of the mitigating factors in the treatment response.

DETAILED DESCRIPTION:
Treatment induced neuropathy of diabetes (TIND), also referred to as insulin neuritis, is thought to be a rare iatrogenic cause of neuropathy that occurs in the setting of rapid glycemic control in individuals with a history of prolonged hyperglycemia.

In a recent paper, the investigators reported that a systematic review of all patients seen in a tertiary diabetic neuropathy referral center resulted in the diagnosis of TIND in >10% of patients seen over a 5 year period of time. These individuals developed symptoms of neuropathy as a consequence of a sudden improvement in glycemic control. The neuropathy associated with TIND is a painful small fiber and autonomic neuropathy of acute onset, but is also associated with the simultaneous development of retinopathy and nephropathy.

TIND differs from the most prevalent generalized neuropathy of diabetes, the distal sensory-motor polyneuropathy, in several respects. The neuropathic pain has an acute onset, appearing within 8 weeks of glycemic change in contrast to the more insidious onset in the Diabetic sensorimotor polyneuropathy (DSP). The pain in TIND is more severe, and poorly responsive to interventions including opioids, whereas most patients with DSP respond to non-opioid interventions. Although the distribution of the pain is length dependent in individuals with TIND, it is frequently far more extensive than in DSP and the associated allodynia and hyperalgesia are much more prevalent. Autonomic symptoms and signs are common, prominent and appear acutely, in contrast to the relatively lower prevalence, gradual onset and slow progression in DSP. Finally, both the pain and autonomic features may be reversible in some patients.

The pathogenic mechanisms whereby this change in glucose results in nerve damage and/or dysfunction are not known. Proposed mechanisms include endoneurial ischemia due to epineurial arterio-venous shunts, apoptosis due to glucose deprivation, microvascular neuronal damage due to recurrent hypoglycemia and ectopic firing of regenerating axon sprouts, but these possibilities are unproven. A potential role for inflammation as a cause of TIND is supported by studies showing an increase in pro-inflammatory cytokines provoked by experimental hypoglycemia. This is reinforced by the association of hyperalgesia with prior exposure to hypoglycemia.

Other microvascular complications are commonly seen in patients with TIND. The simultaneous development of TIND, retinopathy and nephropathy in our cohort suggests a common systemic mechanism likely resulting in microvascular disease. Prior reports of 'early worsening retinopathy' associate a greater risk of retinopathy development with every percentage point decrease in the glycosylated hemoglobin, a result that parallels the neuropathy development in TIND. Furthermore, a link between hypoglycemia, production in pro-inflammatory cytokines, and the development of retinopathy has been proposed.

Treatment induced neuropathy is an iatrogenic cause of an acute, painful autonomic neuropathy in patients with poor glycemic control. Although the underlying mechanism is not yet known, there is a clear relationship between a rapid rate of glycemic control and the development of microvascular complications. Our preliminary data on upregulation of cytokines in individuals with TIND, and the similar findings noted in early worsening retinopathy, suggest the possibility that early intervention may improve outcomes.

The investigators have studied over 100 individuals with TIND in a longitudinal fashion. The characteristic disease progression is well described and related to the magnitude of the change in HbA1c. All patients develop severe neuropathic pain and progressive small fiber and autonomic neuropathy. The neuropathy progresses over 18-24 months and then may gradually improve.

The investigators have studied 4 patients with TIND that developed the acute onset of autonomic and peripheral neuropathy in the setting of rapid glycemic control. All 4 individuals had regular detailed neurological examinations, skin biopsy analysis of nerve fiber density, autonomic function testing and retinal examinations.

Within 4 weeks of the onset of neuropathic pain (within 8 weeks of the change in glucose levels), they were offered a trial of immune globulin administration at a dose of 2grams/kg divided into 5 doses of 0.4 grams/kg for 5 days. In 3 of 4 patients there was significant improvement in neuropathic pain (>50%) and autonomic dysfunction with 4 weeks of immune globulin administration. In addition, there was a clinically significant increase in intra-epidermal nerve fiber density after 6 months (findings not seen in the large cohort of individuals that were untreated). One patient did not exhibit any clear improvement in neuropathic pain or autonomic dysfunction. Prior to immune globulin administration the investigators measured circulating cytokine levels in these 4 individuals. Those that responded tended to have higher circulating cytokine levels than that the individual that did not.

The investigators propose a prospective therapeutic study to determine the efficacy of IVIG in improving both neuropathic pain and nerve fiber structure and function in individuals with TIND. In addition, the investigators will attempt to define mechanisms that will predict success in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of diabetes and treatment induced neuropathy (defined by the onset of neuropathic pain and signs of small fiber or autonomic neuropathy within 8 weeks of a change in HbA1C exceeding 3 points over 3 months).
* Ages 18-60.
* BMI ≤ 30.
* Nonsmoker.
* Consumption of up to 4 alcoholic beverages per week.
* No history of substance abuse or dependence with 1 year prior to screening.
* Normal ECG.
* Vital Signs within normal range (with the exception of a resting tachycardia which is expected in all subjects due to neuropathic pain; research subjects with a heart rate greater than 110 bpm, however, will be excluded).
* CBC, standard chemistry panel within normal limits.
* Standard coagulation studies (within BIDMC laboratory normal limits) including PT, PTT, platelets.
* D-dimer <0.05 FEU.

Exclusion Criteria:

* Female subjects of childbearing potential with a positive urine pregnancy test.
* BMI >30.
* No other known cause of neuropathy (chemotherapy, toxins, other medical disorder - all subjects have diabetes so this would not be an exclusionary factor).
* Anticoagulation with warfarin, aspirin & Plavix together or other anticoagulant that would place subjects at undue risk of bleeding from a skin biopsy. Aspirin or Plavix alone are not an exclusion criterion.
* Clinically active coronary artery or cerebrovascular disease.
* Cardiac insufficiency (NYHA Grade III-IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable advanced ischemic heart disease.
* History of congenital or acquired coagulopathy or thromboembolic disease before the age of 55 or arterial thromboembolic disease before the age of 45.
* History of Deep Venous Thrombosis (DVT) and/or Pulmonary Embolism (PE).
* Evidence of lower extremity deep vein thrombosis at screening including limb swelling, pain or discoloration and or risk of thrombotic event as assessed by Wells criteria.
* Known history of blood hyperviscosity.
* Evidence of severe vascular disease (history of ulceration, poor wound healing, vascular claudication).
* History of allergic reaction to local anesthesia for skin biopsies or history of scarring or keloid formation.
* History of renal dysfunction that includes glomerular filtration rate <60 mL/min, or creatinine of >2.0 mg/dL.
* Known IGA deficiency with antibodies to IgA.
* History of hypersensitivity, anaphylaxis or severe systemic response to immunoglobulin, blood or plasma derived products.
* Positive Direct Antiglobulin Test (DAT) prior to administration or history of hemolytic anemia.
* Subject who is unlikely to comply with the study protocol, or in the opinion of the investigator, would not be a suitable candidate for participation in the study.

Criteria for discontinuation:

* Pregnancy: women of childbearing potential will have a urine pregnancy test at every visit. Subjects who become pregnant will be discontinued from the study.
* A Grade 3 or higher allergic reaction within 24 hours of IVIG/Placebo infusion.
* Any thromboembolic events (e.g. myocardial infarction, stroke, venous thromboembolism)
* Clinically significant hematologic complications (e.g. hemolysis and/or neutropenia).
* Withdrawal by subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gibbons, MD, Principal Investigator — Beth Israel Deaconess Medical Cednter
Locations (1):
- Beth Israel Deaconness Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bril V. NIS-LL: the primary measurement scale for clinical trial endpoints in diabetic peripheral neuropathy. Eur Neurol. 1999;41 Suppl 1:8-13. doi: 10.1159/000052074. PMID 10023123
- [Background] Chantelau E, Meyer-Schwickerath R, Klabe K. Downregulation of serum IGF-1 for treatment of early worsening of diabetic retinopathy: a long-term follow-up of two cases. Ophthalmologica. 2010;224(4):243-6. doi: 10.1159/000260231. Epub 2009 Nov 24. PMID 19940532
- [Background] Dabby R, Sadeh M, Lampl Y, Gilad R, Watemberg N. Acute painful neuropathy induced by rapid correction of serum glucose levels in diabetic patients. Biomed Pharmacother. 2009 Dec;63(10):707-9. doi: 10.1016/j.biopha.2008.08.011. Epub 2008 Sep 16. PMID 18848759
- [Background] Dotson S, Freeman R, Failing HJ, Adler GK. Hypoglycemia increases serum interleukin-6 levels in healthy men and women. Diabetes Care. 2008 Jun;31(6):1222-3. doi: 10.2337/dc07-2243. Epub 2008 Mar 10. PMID 18332163
- [Background] Freeman R, Baron R, Bouhassira D, Cabrera J, Emir B. Sensory profiles of patients with neuropathic pain based on the neuropathic pain symptoms and signs. Pain. 2014 Feb;155(2):367-376. doi: 10.1016/j.pain.2013.10.023. Epub 2013 Oct 25. PMID 24472518
- [Background] Gibbons C, Freeman R. The evaluation of small fiber function-autonomic and quantitative sensory testing. Neurol Clin. 2004 Aug;22(3):683-702, vii. doi: 10.1016/j.ncl.2004.03.002. PMID 15207880
- [Background] Gibbons CH, Adler GK, Bonyhay I, Freeman R. Experimental hypoglycemia is a human model of stress-induced hyperalgesia. Pain. 2012 Nov;153(11):2204-2209. doi: 10.1016/j.pain.2012.06.030. Epub 2012 Aug 23. PMID 22921261
- [Background] Gibbons CH, Freeman R. Treatment-induced diabetic neuropathy: a reversible painful autonomic neuropathy. Ann Neurol. 2010 Apr;67(4):534-41. doi: 10.1002/ana.21952. PMID 20437589
- [Background] Gibbons CH, Freeman R. Treatment-induced neuropathy of diabetes: an acute, iatrogenic complication of diabetes. Brain. 2015 Jan;138(Pt 1):43-52. doi: 10.1093/brain/awu307. Epub 2014 Nov 11. PMID 25392197
- [Background] Gibbons CH, Illigens BM, Wang N, Freeman R. Quantification of sweat gland innervation: a clinical-pathologic correlation. Neurology. 2009 Apr 28;72(17):1479-86. doi: 10.1212/WNL.0b013e3181a2e8b8. PMID 19398703
- [Background] Early worsening of diabetic retinopathy in the Diabetes Control and Complications Trial. Arch Ophthalmol. 1998 Jul;116(7):874-86. doi: 10.1001/archopht.116.7.874. PMID 9682700
- [Background] Hilton P, Spathis GS, Stanton SL. Transient autonomic and sensory neuropathy in newly diagnosed insulin dependent diabetes mellitus. Br Med J (Clin Res Ed). 1983 Feb 26;286(6366):686. doi: 10.1136/bmj.286.6366.686. No abstract available. PMID 6402206
- [Background] Honma H, Podratz JL, Windebank AJ. Acute glucose deprivation leads to apoptosis in a cell model of acute diabetic neuropathy. J Peripher Nerv Syst. 2003 Jun;8(2):65-74. doi: 10.1046/j.1529-8027.2003.03009.x. PMID 12795710
- [Background] Lauria G, Hsieh ST, Johansson O, Kennedy WR, Leger JM, Mellgren SI, Nolano M, Merkies IS, Polydefkis M, Smith AG, Sommer C, Valls-Sole J; European Federation of Neurological Societies; Peripheral Nerve Society. European Federation of Neurological Societies/Peripheral Nerve Society Guideline on the use of skin biopsy in the diagnosis of small fiber neuropathy. Report of a joint task force of the European Federation of Neurological Societies and the Peripheral Nerve Society. Eur J Neurol. 2010 Jul;17(7):903-12, e44-9. doi: 10.1111/j.1468-1331.2010.03023.x. PMID 20642627
- [Background] Ohshima J, Nukada H. Hypoglycaemic neuropathy: microvascular changes due to recurrent hypoglycaemic episodes in rat sciatic nerve. Brain Res. 2002 Aug 23;947(1):84-9. doi: 10.1016/s0006-8993(02)02910-4. PMID 12144856
- [Background] Razavi Nematollahi L, Kitabchi AE, Stentz FB, Wan JY, Larijani BA, Tehrani MM, Gozashti MH, Omidfar K, Taheri E. Proinflammatory cytokines in response to insulin-induced hypoglycemic stress in healthy subjects. Metabolism. 2009 Apr;58(4):443-8. doi: 10.1016/j.metabol.2008.10.018. PMID 19303962
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Tesfaye S, Malik R, Harris N, Jakubowski JJ, Mody C, Rennie IG, Ward JD. Arterio-venous shunting and proliferating new vessels in acute painful neuropathy of rapid glycaemic control (insulin neuritis). Diabetologia. 1996 Mar;39(3):329-35. doi: 10.1007/BF00418349. PMID 8721779
- [Background] Tesfaye S, Vileikyte L, Rayman G, Sindrup SH, Perkins BA, Baconja M, Vinik AI, Boulton AJ; Toronto Expert Panel on Diabetic Neuropathy. Painful diabetic peripheral neuropathy: consensus recommendations on diagnosis, assessment and management. Diabetes Metab Res Rev. 2011 Oct;27(7):629-38. doi: 10.1002/dmrr.1225. PMID 21695762
- [Background] Veves A, Backonja M, Malik RA. Painful diabetic neuropathy: epidemiology, natural history, early diagnosis, and treatment options. Pain Med. 2008 Sep;9(6):660-74. doi: 10.1111/j.1526-4637.2007.00347.x. PMID 18828198
- [Background] Wang N, Gibbons CH. Skin biopsies in the assessment of the autonomic nervous system. Handb Clin Neurol. 2013;117:371-8. doi: 10.1016/B978-0-444-53491-0.00030-4. PMID 24095140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride | IGIV-C
Started | 6 | 7
Completed | 3 | 5
Not Completed | 3 | 2
Not completed — Covid | 3 | 2

BASELINE CHARACTERISTICS:
Population: A total of 13 participants were enrolled before COVID-19 pandemic shut down research activities. A total of 8 participants were able to complete the study, 5 stopped mid-study due to the COVID shutdown.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride | IGIV-C | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.5) | 39 (13.3) | 40 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Sensory Neuropathy as Measured by the Utah Early Neuropathy Score (UENS).
Description: The Utah Early Neuropathy Scale (UENS) was developed specifically to detect and quantify early small-fiber sensory neuropathy and to recognize modest changes in sensory severity and distribution.
  The UENS scale ranges from 0 (no neuropathy) to 42 (severe small fiber neuropathy). The outcome measure is the UENS score from 7 weeks (final evaluation) minus the UENS score from the baseline visit. A positive value indicates that neuropathy worsened over the course of the trial (a worse outcome), a negative score indicates that neuropathy improved over the course of the trial (a better outcome).
Time Frame: 7 weeks after first infusion.
Population: A total of 3 participants completed treatment with placebo and 4 with IVIG. The remaining participants were unable to continue due to COVID 19 pandemic shutdown of all research activities. Funding was withdrawn at that time and no further studies were completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.9% Sodium Chloride | IGIV-C
Number analyzed (Participants) | 3 | 4
units on a scale | -1.5 (10.7) | -3.9 (12.4)

2. Primary Outcome: Change in Neuropathic Pain Severity as Measured by the Pain Visual Analogue Scores (VAS).
Description: The visual analog scale (VAS) of pain allows for quantification of neuropathic pain.
  The VAS pain scale is a line with markings that range from 0 (no pain) to 10 (worse pain), with whole digit intervals (thus an 11 point scale).
  This outcome measure is the VAS pain score at the final visit (7 weeks after first infusion) minus the VAS pain score at the baseline visit. A positive result indicates that pain increased over the course of the study (a worse outcome), a negative result indicates that pain improved over the course of the trial (a better outcome).
Time Frame: 7 weeks after first infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.9% Sodium Chloride | IGIV-C
Number analyzed (Participants) | 3 | 4
units on a scale | -1.1 (2.2) | -1.6 (2.4)

3. Secondary Outcome: Change in Neuropathy Severity as Measured by Skin Biopsies.
Description: Skin biopsies will be evaluated by measuring the Intra-epidermal nerve fiber density.
  Nerve fiber density is measured in the number of nerve fibers per millimeter. This outcome measure is the nerve fiber density at the final visit (7 weeks after the initial infusion) minus the nerve fiber density from the baseline visit. A positive result indicates that nerve fiber density increased over the course of the study (a better outcome), a negative result indicates that nerve fiber density decreased over the course of the trial (a worse outcome).
Time Frame: 7 weeks after first infusion
Population: The change in nerve fiber density.
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | 0.9% Sodium Chloride | IGIV-C
Number analyzed (Participants) | 3 | 4
fibers/mm | -0.6 (2.5) | -0.3 (2.3)

4. Secondary Outcome: Change in Autonomic Neuropathy as Measured by Standardized Autonomic Nervous System Testing.
Description: The standardized autonomic nervous system testing evaluates the heart rate variability to paced breathing.
  Heart rate variability is reported in beats per minutes. The outcome measure is the heart rate variability at the final visit (7 weeks after initial infusion) minus the heart rate variability of the baseline visit. A positive result indicates an increase in heart rate variability (a better outcome), a negative result indicates a decrease in heart rate variability (a worse outcome).
Time Frame: 7 weeks after first infusion
Population: A change in the heart rate variability during paced breathing.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | 0.9% Sodium Chloride | IGIV-C
Number analyzed (Participants) | 3 | 4
beats/minute | 2.1 (3.2) | 2.5 (3.4)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Adverse events recorded at the time of infusion, during interim visits and on phone screens between visits.
Arm/Group | 0.9% Sodium Chloride | IGIV-C
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/3 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.9% Sodium Chloride (N=3) | IGIV-C (N=4)
Infusion reactions (General disorders) | 1 (1) | 2 (2) — Chills, fatigue or mild headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02915263/Prot_SAP_001.pdf